CLINICAL TRIAL: NCT05588323
Title: A Phase 1/2, Multicentre, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Naldemedine in Paediatric Patients Who Are Receiving or Who Are About to Receive Treatment With Opioids
Brief Title: Safety and Pharmacokinetics Study of Naldemedine in Paediatric Participants Receiving Opioids
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1907V921F; 2019-003577-25 (EudraCT Number)
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Opioid-Induced Constipation (OIC)
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naldemedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: ≥ 12 to < 18 Years (Experimental): Participants will receive 0.05 milligrams (mg) to 0.2 mg naldemedine based on their body weight once daily for 7 days.
  Interventions: Drug: Naldemedine
- Cohort 2: ≥ 6 to < 12 Years (Experimental): Participants will receive 0.05 mg to 0.2 mg naldemedine based on their body weight once daily for 7 days.
  Interventions: Drug: Naldemedine
- Cohort 3: ≥ 2 to < 6 Years (Experimental): Participants will be enrolled in this cohort after the safety and PK data has been evaluated for cohorts 1 and 2.
  Participants will receive 0.05 mg to 0.2 mg naldemedine based on their body weight once daily for 7 days.
  Interventions: Drug: Naldemedine

INTERVENTIONS:
Drug: Naldemedine — Administered as an oral tablet (0.2 mg dose level only), or oral suspension (all dose levels)
  Other Names: Rizmoic

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic (PK) profile of naldemedine and nor-naldemedine after a single oral dose of naldemedine in pediatric participants who are receiving or about to receive opioids.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

* Participants with cancer or non-cancer pain who are receiving (or who are about to receive) acute or chronic treatment with opioids.
* Participants with either newly diagnosed constipation, a history of constipation treated with laxatives, or are expected to develop constipation after opioid treatment.
* Able to remain in the clinic for blood sampling for at least 12 hours following the first study intervention dose and are able to return for blood sampling at the 24-hour time point.

Weight

* Body mass index within approximately the 3rd to 97th percentile for their age according to the World Health Organization Child Growth Standards.

Exclusion Criteria:

Medical Conditions

* History of a gastrointestinal (GI) neoplasm or an ongoing GI-related issue or any recent (within last 1 year) or planned GI tract surgery.
* Signs or symptoms of GI obstruction or participants with recurrent obstruction who may be at increased risk of GI perforation.
* Inability to eat/swallow or have need of a nasogastric tube.
* No bowel movements reported for 7 consecutive days at the time of obtaining informed consent or on the initial day of study intervention administration (Study Day 1).
* History of more than 1 week of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 neutropenia or thrombocytopenia with clinical sequelae.
* Participants who need mechanical ventilation.
* Severe CTCAE Grade 3 or above hepatic or renal impairment including end-stage renal disease requiring hemodialysis, as determined by the investigator.
* Progressive neurological disorders or potential disruption to the blood-brain barrier (for example, primary brain malignancies, central nervous system metastases, active multiple sclerosis, etc.) considering the risk of opioid withdrawal or reduced analgesia.

Prior/Ongoing Medications

* Currently receiving the first cycle of chemotherapy.
* Previously received naldemedine.

Other Exclusions

- Positive pregnancy test for females of childbearing potential.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Time to Achieve Maximum Plasma Concentration (Tmax) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
AUC Extrapolated From Time Zero to Infinity (AUC0-inf) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Terminal Elimination Rate Constant (λz) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Terminal Elimination Half-life (t1/2,z) of Naldemedine and Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Apparent Total Clearance (CL/F) of Naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Mean Residence Time (MRT) of Naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Apparent Volume of Distribution in the Terminal Phase (Vz/F) of Naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Metabolic Ratio of Cmax of Nor-naldemedine to Cmax of Naldemedine (MRM/U, Cmax) for Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose
Metabolic Ratio of AUC of Nor-naldemedine to AUC of Naldemedine (MRM/U, AUC) for Nor-naldemedine | Day 1: 0.5, 1, 5, and 12 hours postdose; Day 2: 24 hours post Day 1 dose, before administering the Day 2 dose; Day 7 (Cohort 1 only): Predose and 1 hour postdose

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 7
Population PK Analysis: Cmax of Naldemedine | Day 1 through Day 7
Population PK Analysis: Tmax of Naldemedine | Day 1 through Day 7
Population PK Analysis: AUC From Time Zero to tau (AUC0-tau) of Naldemedine | Day 1 through Day 7
Population PK Analysis: Accumulation Ratio for Cmax Calculated as Ratio of Day 7 to Day 1 Cmax (RCmax) of Naldemedine | Day 1 through Day 7
Population PK Analysis: Accumulation Ratio for AUC Calculated as Ratio of Day 7 to Day 1 AUC (RAUC) of Naldemedine | Day 1 through Day 7
Palatability of Naldemedine Powder for Oral Suspension in Participants Aged 6 Years and Above | Day 1 through Day 7
  Palatability will be assessed by participant self-reporting using a visual analogue scale (VAS).
Palatability of Naldemedine Powder for Oral Suspension in Participants Aged 2 to Less Than 6 Years | Day 1 through Day 7
  Palatability will be assessed by the investigator or a participant's parent/legal guardian and, if possible, by participant self-reporting using a VAS with facial hedonic scale.
Ability to Swallow Naldemedine Tablets | Day 1 through Day 7
  Ability to swallow will be assessed by self-reported ease of swallowing after the first dose. Willingness to swallow will be assessed based on the participant's behavior indicative of a negative response and the response to the taste of naldemedine powder for oral suspension formulation compared to the participant's response to all other oral medications currently being given.

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (16):
- University Center Mother Theresa , Hospital - Onco-hematology department, Tirana, Albania
- Yeolyan Hematology. , and Oncology Center -, Yerevan, Armenia
- Belgium (3):
  - CHU Saint-Pierre Clinical Trials Unit, Brussels
  - Universitair Ziekenhuis Brussel (UZBrussel) - Department of Anesthesiology and Perioperative Medicine, Brussels
  - University Hospitals Leuven Pediatrisch hemato-oncology, Leuven
- University Clinical Hospital , Mostar, Mostar, Bosnia and Herzegovina
- France (4):
  - Chu de Caen, Caen
  - Hôpital Béclère Service de Pédiatrie Centre de Référence des Maladies Héréditaires du Métabolisme Hépatique (CRMHMH), Clamart
  - Hôpital Jeanne de Flandre Antenne du CIC pédiatrique - Niveau 0 CHU de Lille, Lille
  - Hôpital Armand Trousseau Service Hématologie et Oncologie Pédiatrique, Paris
- Italy (3):
  - Instituto Nazionale dei Tumori, Milan
  - Citta della Salute e della Scienza di Torino, Torino
  - Maternal and Child Health Institute IRCCS Burlo Garofolo, Pain and pediatric palliative care service, Trieste
- National Center for Child Health and Development, Tokyo, Japan
- North Macedonia (2):
  - PHI University Clinic for Children's , Surgery, Skopje
  - University Clinic for Childrens Diseases , Department of Oncology, Hematology and , Malignant Hemopathy, Skopje

IPD SHARING:
Plan to Share IPD: No